CLINICAL TRIAL: NCT02921906
Title: Assessing the Effect of Food Composition on Postprandial Insulin Secretion in KCNJ11 Neonatal Diabetes (FoND Study)
Brief Title: Effect of Food Composition on Postprandial Insulin Secretion in Neonatal Diabetes
Acronym: FoND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R&D no 1701366
Record Dates: First submitted 2016-09-20; First posted 2016-10-03 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Neonatal Diabetes
Keywords: Insulin; Glucose; Incretin; GLP-1; Food
MeSH Terms: conditions — Insulin Resistance | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neonatal diabetes (Experimental): People with neonatal diabetes due to mutations in the KCNJ11 gene who are treated with sulphonylureas and not on insulin.
  Interventions: Other: High protein meal; Other: High carbohydrate meal; Drug: Paracetamol; Other: Fasting state - sulphonylurea only
- Non-diabetic controls (Active Comparator): People without diabetes.
  Interventions: Other: High protein meal; Other: High carbohydrate meal; Drug: Paracetamol
- Controls with Type 2 Diabetes (Active Comparator): People with Type 2 diabetes who are treated with sulphonylurea medication.
  Interventions: Other: High protein meal; Other: High carbohydrate meal; Drug: Paracetamol

INTERVENTIONS:
Other: High protein meal — Breakfast with high protein / low carbohydrate content
Other: High carbohydrate meal — Breakfast with high carbohydrate / low protein content
Drug: Paracetamol — Standard dose of paracetamol administered with each meal to allow measurement of rate of gastric emptying.
  Other Names: Acetaminophen
Other: Fasting state - sulphonylurea only — People with diabetes take sulphonylurea medication in the absence of any food stimulus
  Arms: Neonatal diabetes

SUMMARY:
Neonatal diabetes is diagnosed before 6 months of age and causes high blood glucose levels due to the pancreas not secreting insulin. Neonatal diabetes can be caused by a change in a DNA region called the KCNJ11 gene. KCNJ11 encodes a channel in the pancreas that acts as a switch to turn 'on' and 'off' insulin secretion. A change in KCNJ11 results in a faulty channel, which keeps insulin secretion 'switched off'. The diabetes can be treated with tablets called sulphonylureas that switch the pancreatic channel 'on', allowing it to secrete insulin in response to gut hormones called incretins. Previous research has shown that patients who switch from insulin to sulphonylureas have better blood glucose control, including fewer episodes of hypoglycaemia (glucose dropping too low), and also avoid the need for injections. It is thought that serious side effects from sulphonylureas are uncommon in KCNJ11 neonatal diabetes. Some patients report low glucose after meals and we think this may be because they make too much insulin if they eat a meal with protein but low amounts of carbohydrate. The investigators will test this by giving study participants different meals and measuring the amount of insulin, glucose and incretin hormone in the blood afterwards.

DETAILED DESCRIPTION:
Anecdotal evidence from routine clinical care suggests that patients with sulphonylurea-treated KCNJ11 neonatal diabetes, when they eat, may experience mild hypoglycaemia if the food consumed lacks carbohydrate. It has been suggested that this may be due to regulation of insulin secretion via the incretin pathway as opposed to the classical ATP pathway. Therefore the investigators hypothesise that foods with a relatively high protein content compared to those with a relatively high carbohydrate content will result in excessive insulin secretion and relatively lower glucose values in KCNJ11 patients. This would be in contrast to healthy control subjects or subjects with SU-treated T2D where the insulin secretion will be moderated by the ambient glucose via the classical ATP pathway. The investigators will formally study this hypothesis by comparing the insulin, glucose and incretin hormone responses to a high protein meal with a high carbohydrate meal in people with KCNJ11 neonatal diabetes, people without diabetes and people with sulphonylurea-treated Type 2 Diabetes. To assess whether any effect seen is due to direct stimulation of the beta cell by the sulphonylurea itself, people with KCNJ11 neonatal diabetes will also undergo the same tests in the fasting state, having taken the sulphonylurea in the absence of any food.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥8yrs.
* Willing and able to provide informed consent (adults i.e. participants aged >16 years).
* Willing and able to provide assent and parents willing to provide informed consent (children and young people <16 years).

Exclusion Criteria:

* Age <8yrs.
* Unable/unwilling to provide informed consent (adults).
* Unable/unwilling to provide assent (children) or parents unwilling to provide informed consent.
* Known liver disease or chronic renal impairment (EGFR <60ml/min).

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06; Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Glucose levels | 240 minutes
  Glucose AUC after each meal.
Insulin levels | 240 minutes
  Insulin AUC after each meal.

SECONDARY OUTCOMES:
GLP-1 levels | 240 minutes
  GLP-1 AUC after each meal.
GIP levels | 240 minutes
  GIP AUC after each meal.
Glucagon levels | 240 minutes
  Glucagon AUC after each meal.
Paracetamol levels | 240 minutes
  Rate of change of paracetamol levels after each meal as marker of gastric emptying.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Hattersley, BMBCh DM FRS, Study Chair — University of Exeter
Locations (1):
- Exeter Clinical Research Facility, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bowman P, McDonald TJ, Knight BA, Flanagan SE, Leveridge M, Spaull SR, Shields BM, Hammersley S, Shepherd MH, Andrews RC, Patel KA, Hattersley AT. Patterns of postmeal insulin secretion in individuals with sulfonylurea-treated KCNJ11 neonatal diabetes show predominance of non-KATP-channel pathways. BMJ Open Diabetes Res Care. 2019 Dec 18;7(1):e000721. doi: 10.1136/bmjdrc-2019-000721. eCollection 2019. PMID 31908791